CLINICAL TRIAL: NCT07224139
Title: Sex-specific Risk Factors and Trajectories of Blood Biomarkers for Alzheimer's Disease and Related Dementias
Status: Active, not recruiting | Type: Observational
Sponsor: Anne Murray (Other)
Responsible Party: Sponsor-Investigator, Anne Murray, MD, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Other Study IDs: 1RF1AG079397 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Dementia; Cognitive Dysfunction
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Blood-based ADRD biomarkers show tremendous promise as a non-invasive method to predict and diagnose ADRD. We will measure changes in these biomarkers to determine whether their ability to predict ADRD differs by sex or by other characteristics, and develop a sex-specific ADRD risk score for personalized medicine and clinical trials.

DETAILED DESCRIPTION:
Late-life Alzheimer's disease and related dementias (ADRD) are devastating multifactorial conditions and the major contributors to loss of independence in older age. There is a critical unmet need to identify which individuals are at the great risk of these conditions, thus permitting accurate prognosis and timely preventative interventions to reduce the burden. Yet, while a number of risk factors have been identified for these conditions, sex differences in these associations have rarely been considered. Furthermore, exciting recent advances in blood amyloid, tau and neurodegeneration (AT(N)) biomarkers for ADRD means that they could soon be used as powerful clinical diagnostic and prognostic tools in a personalized medicine approach. However, a number of critical knowledge gaps remain. Importantly, 1) these biomarkers have not been sufficiently examined in longitudinal studies of older community- based populations without diagnosed dementia; 2) it is unclear how participant characteristics such as comorbidities affect the clinical interpretation of these biomarkers; and 3) how their interpretation may differ between men and women. Together, these large knowledge gaps highlight a crucial need to develop the first sex-specific risk score for ADRD that incorporates blood AT(N) biomarkers and ADRD risk factors.

ELIGIBILITY:
Inclusion Criteria:

We will use de-identified data and biospecimens originally collected for a large binational NIA-funded ASPirin in Reducing Events in the Elderly (ASPREE) randomized clinical trial and ongoing observational follow-up (U19 AG062682) for analysis.

Exclusion Criteria:

None

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The data and biospecimens collected for a large-scale study of initially healthy individuals aged 65-98 years from the US and Australia (12,716 whites, 412 blacks, 339 other minorities) with comprehensive annual in-person cognitive assessments, adjudicated clinical outcomes, detailed data on socio-economic status, lifestyle and health factors collected over a median 9+ years, and existing genetic data (APOE4, dementia polygenic risk scores).
Sampling Method: Non-Probability Sample
Enrollment: 13435 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To prospectively measure plasma AT(N) biomarkers and to identify participant characteristics that are associated with these levels separately in women and men. | In a community population of 21,000 older persons without dementia, we will measure changes in these biomarkers over 7 to 10 years
  We hypothesize that:
  1a. There will be sex differences in the cross-sectional biomarker levels, and in their trajectories over time.
  1b. Chronic comorbidities and genetic risk factors (APOE ε4, polygenic risk score) will be associated with 'worse' AT(N) biomarker levels (reflecting worse ADRD pathology) at baseline and with a greater increase over time over time, and that these associations will differ between men and women.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Murray, MD, MSc, Principal Investigator — Hennepin Healthcare Research Institute
Locations (5):
- United States (4):
  - Foundation for Atlanta Veterans Education and Research, Inc., Decatur, Georgia
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - Regents of the University of Minnesota - Advanced Research & Diagnostic, Minneapolis, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
- Monash University, Melbourne, Victoria, Australia